CLINICAL TRIAL: NCT04315675
Title: A Pilot Study to Improve Functional Health Health Status in Minority Women Living With HIV
Brief Title: Improve Functional Health Status in Minority Women With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seton Hall University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SetonHallU
Record Dates: First submitted 2020-02-28; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: HIV/AIDS
Keywords: Promoting functional health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a quantitative intervention study that tests and compares outcomes of three interventions and a control group. The subjects are randomly assigned to one of four study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Guided Imagery Intervention (Experimental): Participants randomly assigned to this group will be provided with a MP3 Player which will have three guided imagery programs The Guided Imagery Programs include: 1.) Relaxation and Wellness; 2.) Immune System Imagery; and 3.) Healing Trauma.
  Interventions: Behavioral: Guided Imagery Intervention
- Cognitive Power Intervention (Experimental): The participant who is randomly assigned to this group completes The Power as Knowing Participation in Change Version II (PKPCT) to determine 1.) Freedom to Act Intentionally, 2.) Involvement in Creating Change, 3.) Freedom to Act Intentionally and 4.) My Involvement in Creating Change.
  Interventions: Behavioral: Cognitive Power Intervention
- Cognitive Power Intervention and Guided Imagery (Experimental): The participant is randomly assigned to this group completes both the Guided Imagery Intervention and the Cognitive Power Intervention.
  Interventions: Behavioral: Combined Guided Imagery and Cognitive Power Intervention
- Control Group (No Intervention): The participant is randomized to the control group and completes all study measures twenty-one days after the baseline data are competed. .

INTERVENTIONS:
Behavioral: Guided Imagery Intervention — The participant listens to a selected Guided Imagery for 21 consecutive days.
  Arms: Guided Imagery Intervention
Behavioral: Cognitive Power Intervention — The participant develops a plan to achieve healthy outcomes and reviews plan for 21 consecutive days.
  Arms: Cognitive Power Intervention
Behavioral: Combined Guided Imagery and Cognitive Power Intervention — The participant completes 21 days of selected Guided Imagery in combination with the development of a plan to achieve healthy outcomes and reviews the plan for 21 days.
  Arms: Cognitive Power Intervention and Guided Imagery

SUMMARY:
HIV is no longer a death sentence, and with adherence to Rapid High Activity Antiretroviral (HAART) protocol women with HIV can achieve a normal life expectancy. In New Jersey there are 11,724 (32.9%) women living with HIV with Essex county in the lead, and they come they come from lowest social strata and educational level and are often single mothers. The purpose of this study is test three study interventions: a cognitive health promotion intervention, a guided imagery intervention and combination of both interventions.

The Significance of the study is to improve the functional health and protocol adherence, to better enable women with HIV to achieve a normal life expectancy. The Methodology is an intervention study that uses a classic four group pretest post-test experimental design with random assignment, and the subjects for the study will be 80 women living with HIV. The interventions will be delivered within a three-week time frame followed by post testing at the end of the third week in Newark,New Jersey. The results of this study will be used as preliminary data to support a grant proposal to be submitted to the National Institutes of Health. The Results of this study are important as they will support improved health function and adherence to treatment protocols for marginalized poor women with HIV to achieve outcomes on par with men.

DETAILED DESCRIPTION:
Background: Among the more than one million persons in the United States living with HIV/AIDS, women comprise approximately 25% or 280,000 of persons infected with HIV (CDC, 2015). According to The CDC (2015) in 2010 there were 7800 new cases of HIV in women. Black/African American Women accounted for 5,300 of these women, followed by 1200 Hispanic/Latino women who were newly diagnosed with HIV.

The women with HIV/AIDS in the United States largely come disproportionately from minorities who are marginalized at the lowest strata of society with Black and Hispanic inner city women accounting for approximately 80% of all cases.The fourth leading cause of death in Black women, HIV/AIDs is a disease of poor women who count HIV as not the main problem, but one of more than a dozen life challenges that they encounter in their day to day living. (Hansell, Hughes, Caliandro, Budin,1999). HIV in women affects the entire family especially the children of these women who lead a highly deprived and compromised life. The day to day challenges that these women encounter to stay alive causes them to struggle to maintain their own health with quality lives and to adequately provide for their children. By comparison men with HIV tend to come from a higher social stratum have a higher level of educational and professional attainment. The current treatment for HIV/AIDS is High Activity Antiretroviral therapy (HAART) which provides a simple one pill regimen taken daily. This HIV regimen is highly effective in reducing viral load and an increasing CD4 counts. The HIV disease process is effectively managed by HAART and mitigates the progression of disease thus rendering it a chronic disease state. With the effective management of HIV, it is critical for the person to adhere to the HAART Protocol, as well as manage one's own health status through a better understanding of health promotion and disease prevention. Purpose: The purpose of this study is to test interventions for women with HIV/AIDS aimed at improving their functional health status and protocol adherence by promoting positive health behaviors enabling them to achieve higher functional health. These results will be used as preliminary data for an NIH grant proposal for a large-scale intervention study on the HAART protocol adherence and the functional health of women with HIV/AIDS.

Specific Aims:

The Specific aims for this study are focused on women living with HIV are as follows:

1. To describe patterns of health, wellness, protocol adherence CD4 counts, viral load and Functional Health Status.
2. To test the effect of a guided imagery intervention on HAART Adherence, Viral load, CD4 Counts and Functional Health Status.
3. To test the effect of a cognitive power intervention on HAART Adherence, Viral load, CD4 Counts and Functional Health and Functional Health Status..
4. To test the effect of a combined guided imagery intervention in combination with Cognitive Power Intervention on HAART adherence, Viral Load, CD4 Counts and Functional Health Status

The outcome variables will be generated by the study measures and will include: CD4 counts; Viral Load; the EF-36v2 Health Survey and the Power as Knowing Participation in Change (PKPCT)Tool.

Significance:Women living with HIV/AIDS are largely from medically under-served communities and are primarily from minority populations. Women living with HIV/AIDS who are adhere to their HIV treatment protocol need to make choices that promote their functional health and prevent co-morbidity which will enable them to lead normal lives and become more productive members of society.

Conceptual Framework: Barrett's Power as Knowing Participation in Change Theory provides the framework for this study. Barrett "Power is Knowing Participation in Change conveys the notion that power is the capacity to participate knowingly in change which is manifest by awareness, choices, freedom to act intentionally and involvement in creating change. The two types of power are: power as control and power as freedom. The overall focus in this study is to aid subjects to effectively deploy their power to best enable the best possible achievement of improved health function.

Methodology: This study is a quantitative intervention study that tests and compares outcomes of three interventions and a control group. The design is a classic pretest control group design that includes three intervention groups that will be compared to a control group. Within this design subjects are randomly assigned to one of the four study groups:

1. Group One R Pre-test X (Guided Imagery Intervention) Post Test n=20.
2. Group Two R Pre-test Y (Cognitive Power Intervention) Post Test n=20.
3. Group Three R Pre-test XY (Combination Intervention Post Test n=20.
4. Control Group Post Test n=20.

Total Number of Subjects 80

Subjects: Subjects are women with HIV who are compliant on a HAART treatment protocol. With four groups a sample of 80 subjects is projected with 20 subjects per group. Subjects with multi-system or debilitating complications, limited cognitive or language will be excluded from the sample.

Instrumentation/ Study Measures: Background Demographic Questionnaire- baseline data regarding age, sex, marital status, health status, HIV history, Family structure, treatment plan. CD4 counts- CD4 measures CD4 cells that are in a human body. CD4 cells play an important role in the immune system to infection. CD4( Cluster of Differential 4) counts below 200 place an individual at high risk for serious illnesses. The normal CD4 count in HIV sero-negative persons ranges between 460 and 1600. CD4 counts are standard in HAART protocols. Viral Load- Viral load is a blood test that measures how much HIV is in a person's body. Patients on HIV treatment protocol have been tested for viral load. SF-36v2 Health Survey- The Optimum TM SF 36v2 Health Survey asks 36 questions to measure functional health from the patient's perspective. The higher the score the higher the Health Function.The Power as Knowing Participation in Change Tool (PKPCT is based upon the four dimensions of power which are: awareness; choices:freedom to act intentionally and involvement in creating change (Barrett, 2003). Power as knowing participation is being aware of what one is choosing to do, and doing it intentionally. Awareness and freedom to act intentionally guide choices and involvement in creating changes. Power is freedom to make aware choices for life situations including health promoting changes. Free to act as one wishes is critical to power. Awareness is the focusing of attention on what one perceives to exists. Choices are selections from possibilities for participating in experiences Freedom to act intentionally is the experience of one's capacity to do or bring about what one has in mind. Involvement in creating change is innovative engagement in the unpredictable human-environment mutual process to actualize some potential. The score range for each scale is 12-84 and for the total scale 48-336. Lower scores indicate less power and higher scores indicate higher power.

Procedures: After informed consent is obtained, subjects are randomly assigned to one of four study groups. Baseline data are collected and for participants in the intervention groups their assigned intervention begin.

Interventions: Guided Imagery- is an intervention based on the mind body connection whereby thoughts guide the imagination toward a relaxed and focused state. Sessions will be completed for 21 consecutive days beginning at the baseline with measures again repeated 21 days post baseline. The Cognitive Power Intervention on Health Function- The cognitive power intervention on health function uses the subject's power profile to set attainable goals to act intentionally to create specific changes in one's life aimed at the improvement of the participants' Health Function.

Statistical Analysis: The analysis will include both descriptive and multivariate analysis to test for differences between study groups using the .05 level of significance to test for differences.

Results/Outcomes: These results will provide preliminary data for a large scale NIH grant proposal. The study will determine if women living with HIV using study interventions are able to achieve improved health function which ultimately will contribute an improved life expectancy. These results can be useful as a model to improve health function in women with chronic diseases (Diabetes, Cancer Cardiac etc.)

References:

Henry Kaiser Foundation. (2014) Women in HIV AIDS in the United States. New Jersey Department of Health and Human Services. HIV/AIDS among Women in New Jersey, 2016. Statistics Center/HIV/AIDS 2016 and 2017) https//www.cdc.gov.hiv.overview.

ELIGIBILITY:
Inclusion Criteria:

* Women participants diagnosed with HIV
* Must speak and write in English

Exclusion Criteria:

* Women participants with debilitating complications
* Women participants with Cognitive Impairment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with HIV.
Enrollment: 80 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
CD4 Counts | Measured at the baseline
  Cells in human body measure response immune system to infection
CD4 Counts | Measured 21 days after the baseline
  Cells in human body measure response immune system to infection
Viral Load | At the baseline
  Sero blood assessment of amount of HIV virus.
Viral Load | Twenty-one days following the baseline
  Sero blood assessment of amount of HIV virus
SF-36v2 Health Survey | At the baseline
  Functional Health from the participants perspective
SF-36v2 Health Survey | Twenty-one days after the baseline
  Functional Health from the participants perspective
Power as Knowing Participation in Change (PKPCT) | At the Baseline.
  Subjects Power Profile to Create Change
Power as Knowing Participation in Change (PKPCT) | Twenty-one days after the baseline.
  Subjects Power Profile to Create Change

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis S Hansell, EdD, Principal Investigator — Seton Hall University
Locations (1):
- Seton Hall University, College of Nursing, Nutley, New Jersey, United States

REFERENCES:
- [Background] Barrett EA. Power as knowing participation in change: what's new and what's next. Nurs Sci Q. 2010 Jan;23(1):47-54. doi: 10.1177/0894318409353797. PMID 20026728
- [Background] Caroselli C, Barrett EA. A review of the power as knowing participation in change literature. Nurs Sci Q. 1998 Spring;11(1):9-16. doi: 10.1177/089431849801100105. PMID 9555424
- [Background] Hansell PS, Hughes CB, Caliandro G, Russo P, Budin WC, Hartman B, Hernandez OC. The effect of a social support boosting intervention on stress, coping, and social support in caregivers of children with HIV/AIDS. Nurs Res. 1998 Mar-Apr;47(2):79-86. doi: 10.1097/00006199-199803000-00006. PMID 9536191
- [Background] Hansell PS, Hughes CB, Caliandro G, Russo P, Budin WC, Hartman B, Hernandez OC. Boosting social support in caregivers of children with HIV/AIDS. AIDS Patient Care STDS. 1999 May;13(5):297-302. doi: 10.1089/apc.1999.13.297. PMID 10356809